CLINICAL TRIAL: NCT00142727
Title: The Variability of Agonist and Antagonist Effects as a Function of Level of Physical Dependence
Brief Title: Opioid Agonist and Antagonist Effects on Opioid Dependence
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to halt in funding; may resume recruiting in future
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Johns Hopkins University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-08045-6; R01-08045-6; DPMC
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2007-07

CONDITIONS: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Methadone; Analgesics, Opioid; Narcotic Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Methadone
Drug: Full opioid agonist
Drug: Partial opioid agonist
Drug: Opioid antagonist

SUMMARY:
The purpose of this study is to examine the acute agonist and antagonist effects of a full opioid agonist medication, an opioid antagonist medication, and a partial opioid agonist medication in individuals who have different levels of physical opioid dependence.

DETAILED DESCRIPTION:
The pharmacological effects of opioids in opioid dependent individuals can vary as a function of the characteristics of the opioid being studied (e.g., whether it is an agonist, partial agonist, or antagonist; the dose administered; and the route of administration). Another important set of factors influencing the effects produced by opioids is the characteristics of the organism to which the opioid is being administered. One such characteristic is the level of physical dependence in individuals.

Participants in this study will be maintained on different dose levels of an opioid agonist (methadone). The participant will be challenged with a prototypic opioid agonist, antagonist, and a mixed agonist-antagonist with partial agonist features in order to determine the effects that each has on the human body.

ELIGIBILITY:
Inclusion Criteria:

* Active opioid dependence
* Qualifies for opioid agonist treatment (e.g., methadone or buprenorphine)
* Fulfills DSM-IV diagnostic criteria for opioid dependence

Exclusion Criteria:

* Significant medical problems, including insulin dependent diabetes mellitus
* Non-substance use psychiatric disorders (e.g., schizophrenia)
* Currently seeking treatment for substance abuse

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2004-01; Study Completion 2006-02

PRIMARY OUTCOMES:
Opiate withdrawal | up to one day
Opiate agonist symptoms | up to one day
Physiologic measures | up to one day

CONTACTS AND LOCATIONS:
Overall Officials: Eric C. Strain, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University (BPRU) Bayview Campus, Baltimore, Maryland, United States